CLINICAL TRIAL: NCT02730702
Title: Colon Cancer Risk-stratification Via Optical Analysis of Rectal Ultrastructure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: American BioOptics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ABO 2016-01
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: LEBS - Low coherence enhanced backscattering — Unprepped patients will have the LEBS probe brought into contact with the rectal mucosa, upon which 10 random readings will be obtained.

SUMMARY:
This is a study whose focus is on understanding the clinical utility of rectal ultrastructure in detecting colonic neoplasm. The method uses Low-coherence Enhanced Backscattering Spectroscopy (LEBS).

DETAILED DESCRIPTION:
The investigators use an optic probe which is a small device that uses light to assess the colon tissue. This probe will be used to identify subjects who do and do not have precancerous changes in the colon by capturing the light reflected back from the rectal wall and that will be assessed without the need for colonoscopy and bowel preparation (i.e unprepped). This device may detect early cancerous changes in colon tissue with higher accuracy than current tests.

ELIGIBILITY:
Inclusion Criteria:

- Subjects are eligible if they were scheduled for colonoscopy for colon cancer screening or surveillance

Exclusion Criteria:

* age <50
* personal/family history of colonic neoplasia
* personal history of coagulopathy
* (retrospectively) failure to complete or inadequate colonoscopy
* any patients harboring non-pathoglocially normal rectum (i.e. presence of lesion, inflammation, polyp, adenomas at rectum)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be obtained in the gastroenterology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Whether rectal LEBS readings can predict the presence of advanced adenomas in the colon. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: The Quyen Nguyen, Ph.D., Principal Investigator — American BioOptics
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will assure the confidentiality of all human subjects' data and will adhere to all HIPAA rules by, for example, de-identifying data as appropriate to ensure compliance with human subject confidentiality requirements. The investigators will share research outcomes through conference presentations, and through publications as soon as is feasible after peer review.

REFERENCES:
- [Background] Radosevich AJ, Mutyal NN, Eshein A, Nguyen TQ, Gould B, Rogers JD, Goldberg MJ, Bianchi LK, Yen EF, Konda V, Rex DK, Van Dam J, Backman V, Roy HK. Rectal Optical Markers for In Vivo Risk Stratification of Premalignant Colorectal Lesions. Clin Cancer Res. 2015 Oct 1;21(19):4347-4355. doi: 10.1158/1078-0432.CCR-15-0136. Epub 2015 May 19. PMID 25991816